CLINICAL TRIAL: NCT01450761
Title: Randomized, Multicenter, Double-Blind, Phase 3 Trial Comparing the Efficacy of Ipilimumab Plus Etoposide/Platinum Versus Etoposide/Platinum in Subjects With Newly Diagnosed Extensive-Stage Disease Small Cell Lung Cancer (ED-SCLC)
Brief Title: Trial in Extensive-Disease Small Cell Lung Cancer (ED-SCLC) Subjects Comparing Ipilimumab Plus Etoposide and Platinum Therapy to Etoposide and Platinum Therapy Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA184-156; 2011-000850-48 (EudraCT Number)
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Ipilimumab; Etoposide; etoposide phosphate; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab+Etoposide+Cisplatin/Carboplatin (Experimental): Ipilimumab: IV solution, Intravenous (IV), 10 mg/kg, Once every 3 weeks for 4 doses, then every 12 weeks, Until progression of disease or unacceptable toxicity, or until the maximum treatment period of 3 years is reached
  Etoposide: IV solution, IV, 100 mg/m2, Days 1-3 every 3 weeks, 4 cycles
  Cisplatin: IV solution, IV, 75 mg/m2, Once every 3 weeks, 4 doses
  Carboplatin: IV Solution, IV, Area Under the Curve (AUC) 5, Once every 3 weeks, 4 doses
  Interventions: Biological: Ipilimumab; Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin
- Placebo matching Ipilimumab+Etoposide+Cisplatin/Carboplatin (Placebo Comparator): Placebo matching Ipilimumab: IV solution, IV, 0 mg/kg, Once every 3 weeks for 4 doses, then every 12 weeks, Until progression of disease or unacceptable toxicity, or until the maximum treatment period of 3 years is reached
  Etoposide: IV solution, IV, 100 mg/m2, Days 1-3 every 3 weeks, 4 cycles
  Cisplatin: IV solution, IV, 75 mg/m2, Once every 3 weeks, 4 doses
  Carboplatin: IV Solution, IV, Area Under the Curve (AUC) 5, Once every 3 weeks, 4 doses
  Interventions: Biological: Placebo matching Ipilimumab; Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: Ipilimumab
  Other Names: Yervoy; BMS-734016
  Arms: Ipilimumab+Etoposide+Cisplatin/Carboplatin
Biological: Placebo matching Ipilimumab
  Arms: Placebo matching Ipilimumab+Etoposide+Cisplatin/Carboplatin
Drug: Etoposide
  Other Names: Etopophos; Neoposid; Eposin
Drug: Cisplatin
  Other Names: Platinol
Drug: Carboplatin
  Other Names: Paraplatin

SUMMARY:
The purpose of the study is to determine whether the addition of Ipilimumab to Etoposide and Platinum therapy will extend the lives of patients with Extensive-Stage Disease Small Cell Lung Cancer (ED-SCLC) more than Etoposide and Platinum therapy alone.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Extensive-Stage Disease Small Cell Lung Cancer (ED-SCLC)
* Eastern Cooperative Oncology Group (ECOG) of 0 or 1

Exclusion Criteria:

* Prior systemic therapy for lung cancer
* Symptomatic Central Nervous System (CNS) metastases
* History of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2011-12-13 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (198):
- United States (42):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Sutter Medical Center, Auburn, California
  - UCSD Moores Cancer Center, La Jolla, California
  - University Of Colorado Cancer Center, Aurora, Colorado
  - Florida Cancer Specialists S., Fort Myers, Florida
  - Cancer Specialists, LLC, Jacksonville, Florida
  - Lake City Cancer Care, Lake City, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Medical Oncology, LLC, Augusta, Georgia
  - Quincy Medical Group, Quincy, Illinois
  - Presence Medical Group Hematology Oncology, Skokie, Illinois
  - SIU School Of Medicine, Springfield, Illinois
  - St. Francis Medical Group Oncology And Hematology Specialist, Indianapolis, Indiana
  - Cancer Center Of Kansas, Wichita, Kansas
  - Ashland Bellefonte Cancer Center, Ashland, Kentucky
  - University Of Kentucky, Lexington, Kentucky
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - St Joseph Mercy Hospital, Ypsilanti, Michigan
  - St. Luke'S Cancer Institute, Kansas City, Missouri
  - Southeast Nebraska Hematology & Oncology Consultants, P.C., Lincoln, Nebraska
  - Regional Cancer Care Associates, LLC/Cherry Hill Division, Cherry Hill, New Jersey
  - Memorial Sloan Kettering Nassau, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Hematology Care, Incorporated, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Signal Point Clinical Research Center, Llc, Middletown, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Associated in Oncology and Hematology, Chattanooga, Tennessee
  - The Jones Clinic, PC, Germantown, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - University Of Texas, M. D. Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research And Treatment Center, Lubbock, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Argentina (3):
  - Local Institution, Berazategui, Buenos Aires
  - Local Institution, Buenos Aires
  - Local Institution, Provincia de Sante Fe
- Australia (7):
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Wollongong, New South Wales
  - Local Institution, Chermside, Queensland
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Wodonga, Victoria
  - Local Institution, Perth, Western Australia
- Austria (3):
  - Local Institution, Linz
  - Local Institution, Salzburg
  - Local Institution, Vienna
- Belgium (5):
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Leuven
  - Local Institution, Sint-Niklaas
  - Local Institution, Yvoir
- Brazil (3):
  - Local Institution, Passo Fundo, RS
  - Local Institution, Sao Paulo/SP
  - Local Institution, SP
- Local Institution, Montreal, Quebec, Canada
- Chile (2):
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago
- China (12):
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Harbin, Heilongjiang
  - Local Institution, Wuhan, Hubei
  - Local Institution, Nangjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Xi'an, Shaanxi
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Ürümqi, Xinjiang
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Beijing
  - Local Institution, Shanghai
- Local Institution, Córdoba, Colombia
- Czechia (2):
  - Local Institution, Ostrava - Poruba
  - Local Institution, Prague
- France (4):
  - Local Institution, Caen
  - Local Institution, Rennes
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (15):
  - Local Institution, Bad Berka
  - Local Institution, Bochum
  - Local Institution, Dresden
  - Local Institution, Erlangen
  - Local Institution, Frankfurt am Main
  - Local Institution, Gauting
  - Local Institution, Großhansdorf
  - Local Institution, Hamburg
  - Local Institution, Heidelberg
  - Local Institution, Kassel
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, München
  - Local Institution, Oldenburg
  - Local Institution, Ulm
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, Kowloon
- Hungary (6):
  - Local Institution, Budapest
  - Local Institution, Farkasgyepű
  - Local Institution, Mátraháza
  - Local Institution, Pécs
  - Local Institution, Sopron
  - Local Institution, Szolnok
- Ireland (2):
  - Local Institution, Dublin
  - Local Institution, Limerick
- Israel (5):
  - Local Institution, Beersheba
  - Local Institution, Kfar Saba
  - Local Institution, Petah Tikva
  - Local Institution, Ramat Gan
  - Local Institution, Ẕerifin
- Italy (4):
  - Local Institution, Livorno
  - Local Institution, Lucca
  - Local Institution, Meldola (FC)
  - Local Institution, Siena
- Japan (20):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kashiwa, Chiba
  - Local Institution, Matsuyama, Ehime
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Natori-shi, Miyagi
  - Local Institution, Kurashiki-shi, Okayama-ken
  - Local Institution, Hirakata-shi, Osaka
  - Local Institution, Takatsuki, Osaka
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Ube-shi, Yamaguchi
  - Local Institution, Akashi, Hyogo
  - Local Institution, Fukoka
  - Local Institution, Fukuoka
  - Local Institution, Osaka
  - Local Institution, Oskaka
  - Local Institution, Sendai, Miyagi
  - Local Institution, Tokyo
- Mexico (2):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, San Luis Potosi, S.l.p.
- Netherlands (3):
  - Local Institution, 's-Hertogenbosch
  - Local Institution, Breda
  - Local Institution, Eindhoven
- Peru (2):
  - Local Institution, Cercado
  - Local Institution, Lima
- Poland (7):
  - Local Institution, Elblag
  - Local Institution, Karkow
  - Local Institution, Lublin
  - Local Institution, Otwock
  - Local Institution, Poznan
  - Local Institution, Torun
  - Local Institution, Warsaw
- Portugal (2):
  - Local Institution, Coimbra
  - Local Institution, Lisbon
- Romania (4):
  - Local Institution, Cluj-Napoca, Cluj
  - Local Institution, Craiova, Dolj
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
- Russia (6):
  - Local Institution, Chelyabinsk
  - Local Institution, Krasnodar
  - Local Institution, Kursk
  - Local Institution, Moscow
  - Local Institution, Pyatigorsk
  - Local Institution, Saint Petersburg
- South Africa (3):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Pretoria
- South Korea (5):
  - Local Institution, Goyang-si, Gyeonggji-do
  - Local Institution, Hwasun-eup, Hwasun-gun, Jeollanam-do
  - Local Institution, Busan
  - Local Institution, Seoul
  - Local Institution, Suwon
- Spain (8):
  - Local Institution, A Coruña, Galicia
  - Local Institution, Barcelona
  - Local Institution, Benidorm-alicante
  - Local Institution, Castellon
  - Local Institution, Lleida
  - Local Institution, Majadahonda
  - Local Institution, Málaga
  - Local Institution, Valencia
- Sweden (3):
  - Local Institution, Linköping
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Switzerland (3):
  - Local Institution, Basel
  - Local Institution, Winterthur
  - Local Institution, Zurich
- Taiwan (4):
  - Local Institution, Changhua
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Taoyuan
- Thailand (2):
  - Local Institution, Chiang Mai
  - Local Institution, Songkhla
- United Kingdom (5):
  - Local Institution, Withington, Manchester
  - Local Institution, London
  - Local Institution, Preston
  - Local Institution, Sutton
  - Local Institution, Truro

REFERENCES:
- [Derived] Reck M, Luft A, Szczesna A, Havel L, Kim SW, Akerley W, Pietanza MC, Wu YL, Zielinski C, Thomas M, Felip E, Gold K, Horn L, Aerts J, Nakagawa K, Lorigan P, Pieters A, Kong Sanchez T, Fairchild J, Spigel D. Phase III Randomized Trial of Ipilimumab Plus Etoposide and Platinum Versus Placebo Plus Etoposide and Platinum in Extensive-Stage Small-Cell Lung Cancer. J Clin Oncol. 2016 Nov 1;34(31):3740-3748. doi: 10.1200/JCO.2016.67.6601. PMID 27458307
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1414 enrolled participants, 566 participants each were randomized to Ipilimumab and placebo arms. The remaining 282 participants were not randomized, the most frequently reported reason being that the participants no longer met study criteria.
Groups:
- Ipilimumab and Platinum/Etoposide: During the lead-in chemotherapy (induction) phase, participants received platinum/etoposide (investigator's choice of platinum) every 3 weeks for 4 cycles, with ipilimumab (10 mg/kg IV) every 3 weeks for cycles 3-6. During the treatment with blinded study therapy phase, ipilimumab (10 mg/kg IV) was administered every 12 weeks, beginning 9-12 weeks after the last induction dose, for a maximum treatment period of 3 years from the first dose of ipilimumab.
- Placebo and Platinum/Etoposide: During the lead-in chemotherapy (induction) phase, participants received platinum/etoposide (investigator's choice of platinum) every 3 weeks for 4 cycles, with placebo every 3 weeks for cycles 3-6. During the treatment with blinded study therapy phase, placebo was administered every 12 weeks, beginning 9-12 weeks after the last induction dose, for a maximum treatment period of 3 years from the first dose of placebo.
Period: Randomization
Arm/Group | Ipilimumab and Platinum/Etoposide | Placebo and Platinum/Etoposide
Started | 566 | 566
Completed | 562 | 561
Not Completed | 4 | 5
Not completed — Subject no longer meets study criteria | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Disease progression | 0 | 2
Not completed — Adverse Event unrelated to study drug | 1 | 0
Not completed — Other | 0 | 1
Period: Lead-in Chemotherapy
Arm/Group | Ipilimumab and Platinum/Etoposide | Placebo and Platinum/Etoposide
Started | 562 | 561
Completed | 478 | 476
Not Completed | 84 | 85
Not completed — Disease progression | 33 | 32
Not completed — Adverse event unrelated to study drug | 21 | 19
Not completed — Withdrawal by Subject | 14 | 12
Not completed — Study drug toxicity | 6 | 10
Not completed — No longer meets study criteria | 3 | 7
Not completed — Death | 3 | 3
Not completed — Other | 2 | 2
Not completed — Lost to Follow-up | 2 | 0
Period: Treatment With Blinded Study Therapy
Arm/Group | Ipilimumab and Platinum/Etoposide | Placebo and Platinum/Etoposide
Started | 478 | 476
Completed (Completed = remaining on study therapy) | 0 | 0
Not Completed | 478 | 476
Not completed — Disease progression | 318 | 415
Not completed — Study drug toxicity | 87 | 9
Not completed — Adverse event unrelated to study drug | 27 | 19
Not completed — Subject request to discontinue treatment | 15 | 8
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Death | 5 | 6
Not completed — Other/Unspecified | 5 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Maximum clinical benefit | 1 | 2
Not completed — No longer meets study criteria | 1 | 2
Not completed — Not reported | 2 | 2
Not completed — Poor/non-compliance | 1 | 0
Not completed — Administrative reason by sponsor | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of blinded study therapy
Groups:
- Ipilimumab and Platinum/Etoposide: Participants received platinum/etoposide (investigator's choice of platinum) every 3 weeks for 4 cycles with ipilimumab (10 mg/kg IV) every 3 weeks from cycle 3-6 of Induction phase. During the maintenance phase, ipilimumab (10 mg/kg IV) was administered every 12 weeks, beginning 9-12 weeks after the last induction dose, for a maximum treatment period of 3 years from the first dose of ipilimumab.
- Placebo and Platinum/Etoposide: Participants received platinum/etoposide (investigator's choice of platinum) every 3 weeks for 4 cycles with placebo every 3 weeks from cycle 3-6 during the Induction phase. During the maintenance phase, placebo was administered every 12 weeks, beginning 9-12 weeks after the last Induction dose, for a maximum treatment period of 3 years from the first dose of placebo.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab and Platinum/Etoposide | Placebo and Platinum/Etoposide | Total
Number analyzed (Participants) | 478 | 476 | 954
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.90) | 62.6 (8.61) | 61.9 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 150 | 311
  Male | 317 | 326 | 643

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants Who Received at Least One Dose of Blinded Study Therapy
Description: Overall Survival was defined as the time from the date of randomization until the date of death from any cause. For participants without documentation of death, OS was censored on the last date the participant was known to be alive.
Time Frame: Randomization until date of death, up to March 2015, approximately 38 months
Population: All randomized participants who received at least one dose of blinded study therapy
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ipilimumab and Platinum/Etoposide: Participants received platinum/etoposide (investigator's choice of carboplatin or cisplatin) every 3 weeks for 4 cycles with ipilimumab (10 mg/kg IV) every 3 weeks from cycle 3-6 of Induction phase. During the maintenance phase, ipilimumab (10 mg/kg IV) was administered every 12 weeks, beginning 9-12 weeks after the last induction dose, for a maximum treatment period of 3 years from the first dose of ipilimumab.
- Placebo and Platinum/Etoposide: Participants received platinum/etoposide (investigator's choice of carboplatin or cisplatin) every 3 weeks for 4 cycles with placebo every 3 weeks from cycle 3-6 during the Induction phase. During the maintenance phase, placebo was administered every 12 weeks, beginning 9-12 weeks after the last Induction dose, for a maximum treatment period of 3 years from the first dose of placebo.
Arm/Group | Ipilimumab and Platinum/Etoposide | Placebo and Platinum/Etoposide
Number analyzed (Participants) | 478 | 476
months | 10.97 [10.45 to 11.33] | 10.94 [10.02 to 11.50]
Statistical Analysis 1: Comparison: Ipilimumab and Platinum/Etoposide vs Placebo and Platinum/Etoposide; Test type: Superiority or Other; p = 0.3775, Log Rank; Hazard Ratio (HR) = 0.936, 95% CI 2-sided [0.807 to 1.085] — HR = ipilimumab over placebo

2. Secondary Outcome: Overall Survival in All Randomized Participants
Description: as for outcome 1
Time Frame: From randomization until date of death, up to March 2015, approximately 38 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab and Platinum/Etoposide | Placebo and Platinum/Etoposide
Number analyzed (Participants) | 566 | 566
months | 10.22 [9.59 to 10.81] | 9.95 [9.33 to 10.94]
Statistical Analysis 1: Comparison: Ipilimumab and Platinum/Etoposide vs Placebo and Platinum/Etoposide; Test type: Superiority or Other; p = 0.5678, Log Rank; Hazard Ratio (HR) = 0.961, 95% CI 2-sided [0.838 to 1.102] — HR = ipilimumab over placebo

3. Secondary Outcome: Progression Free Survival (PFS) Time in Participants Who Have Received at Least One Dose of Blinded Study Therapy
Description: Progression-Free Survival was defined as the time from the date of randomization to the date of progression per modified World Health Organization (mWHO) criteria or death, whichever occured first. A participant who died without reported progression per mWHO criteria was considered progressed on the date of death. For those participants who remained alive and did not progress, PFS was censored on the date of last evaluable tumor assessment. For those participants who remained alive and had no recorded post-baseline tumor assessment, PFS was censored on the day of randomization.
Time Frame: From randomization until disease progression, up to March 2015, approximately 38 months
Population: All randomized participants who received at least one dose of blinded study therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab and Platinum/Etoposide | Placebo and Platinum/Etoposide
Number analyzed (Participants) | 478 | 476
months | 4.63 [4.50 to 4.99] | 4.44 [4.37 to 4.63]
Statistical Analysis 1: Comparison: Ipilimumab and Platinum/Etoposide vs Placebo and Platinum/Etoposide; Test type: Superiority or Other; p = 0.0161, Log Rank; Hazard Ratio (HR) = 0.851, 95% CI 2-sided [0.747 to 0.971] — HR = ipilimumab over placebo

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 90 days, up to a maximum of 3 years. Assessed through study completion (May 2017).
Arm/Group | 10 MG/KG IPILIMUMAB + PLATINUM/ETOPOSIDE | PLACEBO + PLATINUM/ETOPOSIDE
Serious Adverse Events (participants affected / at risk) | 316/562 | 278/561
Other Adverse Events (participants affected / at risk) | 519/562 | 520/561
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG IPILIMUMAB + PLATINUM/ETOPOSIDE (N=562) | PLACEBO + PLATINUM/ETOPOSIDE (N=561)
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory distress (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 3
Chest pain (General disorders) | 5 | 5
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Condition aggravated (General disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
General physical condition abnormal (Investigations) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 1
Haematotoxicity (Blood and lymphatic system disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 | 43
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Proctalgia (Gastrointestinal disorders) | 0 | 1
Pyomyositis (Infections and infestations) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 5 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 7
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 2 | 1
Weight decreased (Investigations) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Cardiac tamponade (Cardiac disorders) | 0 | 2
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Death (General disorders) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 42 | 13
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 4 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 13
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 3 | 3
Spinal cord disorder (Nervous system disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Adrenalitis (Infections and infestations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 3
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 3 | 0
Circulatory collapse (Vascular disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Epididymitis (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Full blood count decreased (Investigations) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypophysitis (Endocrine disorders) | 4 | 1
Infection (Infections and infestations) | 3 | 3
Influenza (Infections and infestations) | 2 | 0
Lipase increased (Investigations) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Multi-organ failure (General disorders) | 0 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 3 | 3
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 13
Sudden death (General disorders) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 9
Anxiety (Psychiatric disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 4 | 0
Euthanasia (General disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 5
Neutropenic sepsis (Infections and infestations) | 0 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 6
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Vertebral artery occlusion (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 24 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Disease progression (General disorders) | 6 | 9
Dysphagia (Gastrointestinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1
Embolism (Vascular disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Headache (Nervous system disorders) | 4 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0
Ischaemic neuropathy (Nervous system disorders) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung infection (Infections and infestations) | 1 | 3
Memory impairment (Nervous system disorders) | 0 | 1
Myasthenic syndrome (Nervous system disorders) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pain (General disorders) | 1 | 4
Paraparesis (Nervous system disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0
Pneumonia (Infections and infestations) | 33 | 16
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 14
Right ventricular failure (Cardiac disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Vascular occlusion (Vascular disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Asthenia (General disorders) | 4 | 5
Cellulitis (Infections and infestations) | 0 | 2
Cerebral infarction (Nervous system disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myxoedema (Endocrine disorders) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Sepsis (Infections and infestations) | 7 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Viral infection (Infections and infestations) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 15
General physical health deterioration (General disorders) | 13 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 6 | 7
Partial seizures (Nervous system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 5
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Anaemia (Blood and lymphatic system disorders) | 13 | 23
Ataxia (Nervous system disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 3 | 5
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 4
Device related infection (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Drug hypersensitivity (Immune system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malaise (General disorders) | 1 | 2
Mental status changes (Psychiatric disorders) | 2 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 20
Non-cardiac chest pain (General disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Subileus (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 8
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
H1n1 influenza (Infections and infestations) | 1 | 0
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 | 0
Guillain-barre syndrome (Nervous system disorders) | 1 | 0
Iiird nerve disorder (Nervous system disorders) | 1 | 0
Viith nerve paralysis (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG IPILIMUMAB + PLATINUM/ETOPOSIDE (N=562) | PLACEBO + PLATINUM/ETOPOSIDE (N=561)
Chest pain (General disorders) | 38 | 45
Neutrophil count decreased (Investigations) | 87 | 67
Weight decreased (Investigations) | 46 | 41
Back pain (Musculoskeletal and connective tissue disorders) | 43 | 47
Cough (Respiratory, thoracic and mediastinal disorders) | 94 | 81
Decreased appetite (Metabolism and nutrition disorders) | 169 | 138
Diarrhoea (Gastrointestinal disorders) | 159 | 116
Fatigue (General disorders) | 180 | 170
Hyponatraemia (Metabolism and nutrition disorders) | 53 | 50
Rash (Skin and subcutaneous tissue disorders) | 121 | 28
Abdominal pain upper (Gastrointestinal disorders) | 30 | 24
Haemoglobin decreased (Investigations) | 38 | 32
Hypokalaemia (Metabolism and nutrition disorders) | 47 | 31
Insomnia (Psychiatric disorders) | 53 | 62
Vomiting (Gastrointestinal disorders) | 115 | 97
Alanine aminotransferase increased (Investigations) | 47 | 26
Aspartate aminotransferase increased (Investigations) | 44 | 23
Leukopenia (Blood and lymphatic system disorders) | 73 | 87
Nausea (Gastrointestinal disorders) | 232 | 209
Alopecia (Skin and subcutaneous tissue disorders) | 199 | 208
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 75 | 83
Headache (Nervous system disorders) | 67 | 56
Asthenia (General disorders) | 55 | 61
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 36
Constipation (Gastrointestinal disorders) | 121 | 99
Oedema peripheral (General disorders) | 38 | 27
Pyrexia (General disorders) | 79 | 60
Abdominal pain (Gastrointestinal disorders) | 34 | 33
Anaemia (Blood and lymphatic system disorders) | 171 | 189
Dizziness (Nervous system disorders) | 52 | 59
Hiccups (Respiratory, thoracic and mediastinal disorders) | 26 | 32
Neutropenia (Blood and lymphatic system disorders) | 234 | 261
Platelet count decreased (Investigations) | 39 | 48
Pruritus (Skin and subcutaneous tissue disorders) | 82 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 64 | 84
White blood cell count decreased (Investigations) | 51 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.